CLINICAL TRIAL: NCT06358794
Title: SpermFinder: Machine Learning Based-Personalized Prediction of Sperm Retrieval in Patients With Nonobstructive Azoospermia Prior to Microdissection Testicular Sperm Extraction
Brief Title: Machine Learning Based-Personalized Prediction of Sperm Retrieval Success Rate
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2022692
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Infertility, Male; Azoospermia, Nonobstructive
Keywords: Machine learning; Predictive model; Sperm retrieval
MeSH Terms: conditions — Infertility, Male; Azoospermia, Nonobstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: 2,438 patients diagnosed with NOA were included for model training and validation
  Interventions: Diagnostic Test: Machine learning-based predictive model
- External validation cohort: 174 participants from January 2023 to May 2023 were included as the external validation cohort for online platform

INTERVENTIONS:
Diagnostic Test: Machine learning-based predictive model — The clinical features of participants were used to train, test and validate the machine learning models. Various evaluation metrics including area under the ROC (AUC), accuracy, etc. were used to evaluate the predictive performance of 8 machine learning models.
  Groups: Training cohort

SUMMARY:
Non-obstructive azoospermia (NOA) stands as the most severe form of male infertility. However, due to the diverse nature of testis focal spermatogenesis in NOA patients, accurately assessing the sperm retrieval rate (SRR) becomes challenging. The current study aims to develop and validate a noninvasive evaluation system based on machine learning, which can effectively estimate the SRR for NOA patients. In single-center investigation, NOA patients who underwent microdissection testicular sperm extraction (micro-TESE) were enrolled: (1) 2,438 patients from January 2016 to December 2022, and (2) 174 patients from January 2023 to May 2023 (as an additional validation cohort). The clinical features of participants were used to train, test and validate the machine learning models. Various evaluation metrics including area under the ROC (AUC), accuracy, etc. were used to evaluate the predictive performance of 8 machine learning models.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with nonobstructive azoospermia
* underwent microdissection testicular sperm extraction

Exclusion Criteria:

* without intact clinical information
* low data quality

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nonobstructive azoospermia patients who underwent microdissection testicular sperm extraction at the Reproductive Center of Peking University Third Hospital were respectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2612 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
SRR of micro-TESE | At the time after microdissection testicular sperm extraction
  the sperm retrieval success rate of microdissection testicular sperm extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The raw clinical data are not publicly available. Processed nonsensitive data and analysis code are available from the corresponding author on reasonable request.